CLINICAL TRIAL: NCT02973126
Title: Assessment of Fractional Flow reservE Computed Tomography Versus Single Photon Emission Computed Tomography in the Diagnosis of Hemodynamically Significant Coronary Artery Disease. (AFFECTS)
Brief Title: Heartflow (AFFECTS)
Acronym: AFFECTS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 016-096
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FFRct versus SPECT (Other): Comparison of the diagnostic performance of FFRct and SPECT in subjects with suspected stable CAD
  Interventions: Procedure: FFRct and SPECT

INTERVENTIONS:
Procedure: FFRct and SPECT — enable the comparison of diagnostic performance of FFRct and SPECT in subjects with suspected stable CAD after abnormal SPECT imaging who have no contraindications to coronary computed tomography angiography (CCTA).

SUMMARY:
The overall objective of the AFFECTS Study is to assess agreement between SPECT and FFRct in identifying vessel-specific, hemodynamically significant CAD in patients scheduled for invasive coronary angiography (ICA) based on abnormal SPECT myocardial perfusion scans. In particular, the study will evaluate the ability of FFRct to correctly rule out hemodynamically significant CAD in patients with non-significant CAD or normal coronary arteries who had positive SPECT scans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Providing written informed consent
* Subjects with abnormal SPECT myocardial perfusion imaging results who have been referred for clinically indicated ICA within 90-days of SPECT.
* Ability to undergo cCTA

Exclusion Criteria:

* Acute coronary syndrome (ACS).
* Prior, clinically documented, myocardial infarction (MI).
* Prior coronary artery bypass grafting (CABG)
* Prior coronary stenting
* Evidence of ongoing or active clinical instability including unstable angina, intractable arrhythmia, cardiogenic shock, unstable BP, and severe CHF (NYHA class III or IV) or acute pulmonary edema
* Contraindications for cCTA such as:

  1. Presence of pacemaker or internal defibrillator leads such that coronary visualization is impaired
  2. Chronic atrial fibrillation with uncontrolled ventricular response
  3. Known anaphylactic allergy to iodinated contrast that cannot be pre-medicated
  4. Pregnancy or unknown pregnancy status in women of childbearing age
  5. Contraindication to acute beta blockade
  6. Contraindication to acute sublingual nitrate administration
  7. Prosthetic heart valve such that coronary visualization is impaired
* Contraindications for FFRct such as:

  1. Complex congenital heart disease other than anomalous coronary origins alone
  2. Ventricular septal defect with known Qp/Qs > 1.4
* Requiring an emergent procedure within 48 hours of presentation
* Any active, serious, life-threatening disease with life expectancy less than 2 months
* Inability to comply with study procedures
* Current participation in any other clinical trial involving an investigational device, drug, or dictating care pathways at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Positive finding of hemodynamically significant CAD according to SPECT. | 24 months
Positive finding of hemodynamically significant CAD according to FFRct. | 24 months
Positive finding of hemodynamically significant CAD according to ICA +/- iFFR. | 24 months

SECONDARY OUTCOMES:
Physician intuition regarding presence of vessel-specific, hemodynamically significant CAD after review of FFRct results. | 24 months
Cumulative radiation exposure in the study cohort during SPECT, cCTA, and ICA and potential impact of FFRct in reducing radiation exposure in patients with no hemodynamically significant CAD. | 24 months
Potential economic impact of FFRct in decreasing referral to ICA in patients without hemodynamically significant CAD. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Brown, MD, Principal Investigator — Baylor Research Institute
Locations (1):
- The Heart Hospital Baylor Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No